CLINICAL TRIAL: NCT02419521
Title: A Clinical Evaluation of the Medtronic Resolute Onyx Zotarolimus-Eluting Stent System Medtronic RESOLUTE ONYX Core (2.25 mm - 4.0 mm) Clinical Study
Brief Title: Medtronic RESOLUTE ONYX Core (2.25 mm - 4.0 mm) Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0 - 23Mar2015
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device (Other): Medtronic Resolute Onyx Zotarolimus-Eluting Stent System
  Interventions: Device: Resolute Onyx Stent - 2.25 mm - 4.0 mm

INTERVENTIONS:
Device: Resolute Onyx Stent - 2.25 mm - 4.0 mm

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of the Resolute Onyx Zotarolimus-Eluting Coronary Stent System for the treatment of de novo lesions in native coronary arteries with a reference vessel diameter of 2.25 mm to 4.2 mm.

ELIGIBILITY:
Inclusion Criteria:

* Must be an acceptable candidate for percutaneous coronary intervention (PCI), stenting, and emergent coronary artery bypass graft (CABG) surgery
* Must have clinical evidence of ischemic heart disease, stable or unstable angina, and/or a positive functional study
* Must require treatment of either a) a single target lesion amenable to treatment OR b) two target lesions located in separate target vessels
* Target lesion(s) must be de novo lesion(s) in native coronary artery(ies)

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin and bivalirudin, thienopyridines, cobalt, nickel, platinum, iridium, chromium, molybdenum, polymer coatings (e.g. BioLinx) or a sensitivity to contrast media, which cannot be adequately pre-medicated
* History of an allergic reaction or significant sensitivity to drugs such as zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative
* History of a stroke or transient ischemic attack (TIA) within the prior 6 months
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Concurrent medical condition with a life expectancy of less than 12 months
* Currently participating in an investigational drug or another device trial that has not completed the primary endpoint
* Documented left ventricular ejection fraction (LVEF) < 30% at the most recent evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Price, MD, FACC, FSCAI, Principal Investigator — Scripps Green Hospital
Locations (12):
- United States (12):
  - Scripps Green Hospital, La Jolla, California
  - Morton Plant Hospital, Clearwater, Florida
  - Saint John's Hospital, Springfield, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Saint Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - University Hospitals Elyria Medical Center, Elyria, Ohio
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: Medtronic Resolute Onyx Zotarolimus-Eluting Stent System
  Resolute Onyx Stent - 2.25 mm - 4.0 mm
Period: Overall Study
Arm/Group | Device
Started | 75
Completed | 74
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Device
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 55
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Lumen Loss as Measured by Quantitative Coronary Angiography
Description: In-stent late lumen loss at 8-months post-procedure as measured by quantitative coronary angiography
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Device
Number analyzed (Participants) | 75
mm | 0.24 (0.39)

2. Secondary Outcome: Cardiac Death
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 0

3. Secondary Outcome: Target Vessel Myocardial Infarction (TVMI)
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 2

4. Secondary Outcome: Target Lesion Revascularization (TLR)
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 3

5. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: Defined as death, myocardial infarction (Q wave and non-Q wave), emergent coronary bypass surgery, or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 7

6. Secondary Outcome: Target Lesion Failure (TLF)
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 5

7. Secondary Outcome: Target Vessel Failure (TVF)
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 9

8. Secondary Outcome: Stent Thrombosis (ST)
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 1

9. Secondary Outcome: Cardiac Death and TVMI
Time Frame: 8 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 75
Participants | 2

ADVERSE EVENTS:
Time Frame: All non-serious AEs are collected through the 12 month visit. All serious AEs are collected for the duration of the study.
Arm/Group | Device
Serious Adverse Events (participants affected / at risk) | 27/75
Other Adverse Events (participants affected / at risk) | 66/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=75)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3)
Angina Pectoris (Cardiac disorders) | 2 (2)
Angina Unstable (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 4 (4)
Coronary Artery Perforation (Cardiac disorders) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1)
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Supraventricular Extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 2 (2)
Thyroid Disorder (Endocrine disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 6 (8)
Puncture Site Haemorrhage (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 3 (3)
Cardiac Enzymes Increased (Investigations) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Therapeutic Embolisation (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2)
Shock Haemorrhagic (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=75)
Angina Pectoris (Cardiac disorders) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (7)
Chest Pain (General disorders) | 12 (15)
Fatigue (General disorders) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5)
Cardiac Enzymes Increased (Investigations) | 7 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Dizziness (Nervous system disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Hypertension (Vascular disorders) | 7 (7)
Hypotension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other